CLINICAL TRIAL: NCT01852734
Title: Uterine Fibroid Embolization- Long Term Follow up and Technical Perspectives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Stevo Duvnjak,MD, Medical Doctor, Radiologist, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OUH-2013
Record Dates: First submitted 2013-05-06; First posted 2013-05-14 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Uterine Fibroids; Arterial Embolization
MeSH Terms: conditions — Leiomyoma | interventions — Embolization, Therapeutic; Microspheres

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- embolizations, uterine fibroid (Other): embolization interventions with microspheres
  Interventions: Procedure: embolizations ,uterine fibroid; Procedure: embolizations

INTERVENTIONS:
Procedure: embolizations ,uterine fibroid — 26 patients will be treat with Bead-block microspheres, 500-700 and 700-900µm until flow stop ( " cut the tree" appearance)
  26 patients will be treat with Embosphere, 500-700µm and /or 700-900 until "near stasis " flow stop
Procedure: embolizations — comparison between the two microspheres
  Other Names: microsphere, uterine fibroid

SUMMARY:
The purpose of this prospective non-randomised study is to examine whether two different microspheres (Bead-Block and Embosphere) are equally effective in the treatment of the uterine fibroid controlled with contrast-enhanced MR examination.

Quantitative MR imaging, including dominant fibroid T1, T2 and contrast enhancement characteristics before intervention and 3 months after interventions will be analysed as a potential predictor of volumetric response after embolization.

Another purpose is to determine long-term follow-up in all patient treated in a period from 2001-2011 in OUH analysed retrospectively.

DETAILED DESCRIPTION:
Group 1: 26 patient will be treated with Bead-block microspheres - 700-900 µm microspheres or combinations of one vial 2 ml of 500-700 µm microspheres, follow by 700-900 µm microspheres until blood flow stop ( " cut the tree" appearance).

Group 2: 26 patient will be treated with Embosphere; 500-900 µm until "near-stasis" flow stop in the uterine artery.

Clinical and Technical success will be examined, and radiological follow-up 3 and 12 months after embolization using MR contrast-enhanced examination in a Bead Block group and only 3 months control in Embosphere group to assess total fibroid burden infraction degree and eventually residual contracts fibroid enhancement.

Quantitative MRI dominant fibroid characteristic for and 3 months after an intervention to examine eventually potential of as a possible predictor of the volumetric response of the uterine fibroid.

Retrospective study compromised all patient treated between January 2001 until January 2011 with follow up to January 2014, and re-intervention as well as complications rate analysis.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic uterus fibroma

Exclusion Criteria:

* pelvic infection (cystitis, oophoritis, salpingitis, abscess, urethritis)
* gravidity
* uterus malignancy
* big subserosal fibroma with stalk diameter of <2 cm
* menopausal women
* don,t want to be included into the study

  * concomitant adenomyosis

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2013-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
clinical effect | one year
  Primary goal is to achieve release of symptoms after intervention and it would be compared between the two techniques

SECONDARY OUTCOMES:
reinterventions rate | one year

CONTACTS AND LOCATIONS:
Overall Officials: Stevo Duvnjak, MD, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense, Denmark
  - Odense University Hospital, Odense, Fyn